CLINICAL TRIAL: NCT03739242
Title: A Randomized, Double-blinded, Placebo-controlled, Clinical Study of the Effects of a Nutraceutical Combination on LDL Cholesterol Levels in Subjects With Sub-optimal Blood Cholesterol Levels
Brief Title: Effect of a Treatment With a Nutraceutical Combination on Sub-optimal LDL Cholesterol Levels
Acronym: NATCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A. Menarini Industrie Farmaceutiche Riunite S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEIF/MOF-Col/001
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2018-11

CONDITIONS: Hypercholesterolemia
Keywords: Lipids; Cholesterol; Triglycerides; Dyslipidemia; Low density lipoprotein cholesterol; Dietary Fats; Hyperlipidemias; Dietary Supplements; Food Supplements; Nutraceuticals; Nutriceuticals
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceutical combination (Experimental): One film-coated tablet (1300 mg) per os per day to be taken in the evening. Each tablet contains phytosterols 800 mg, Monascus purpureus (167 mg) titrated at 3% in monacolin K (5 mg), niacin 27 mg, linear aliphatic alcohols titrated to 60% octacosanol.
  Interventions: Dietary Supplement: Nutraceutical combination
- Placebo (Placebo Comparator): One film-coated tablet (1300 mg) per os per day to be taken in the evening. Placebo tablets identical in appearance, size, shape, weight and taste to the active product.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nutraceutical combination — One tablet per os per day to be taken in the evening from randomization (day 0) to the end of the trial (day 56 +/- 3)
  Arms: Nutraceutical combination
Other: Placebo — One tablet per os per day to be taken in the evening from randomization (day 0) to the end of the trial (day 56 +/- 3)
  Arms: Placebo

SUMMARY:
High cholesterol is one of the major controllable risk factor for coronary heart disease. It is well demonstrated that drugs that reduce the intestinal absorption of cholesterol or block the synthesis of cholesterol or the association of both, can reduce cholesterol and reduce rate of cardiovascular events. The trial will evaluate natural alternative to this drug approach testing the effects of a combination of phytosterol, a nutritional that reduce cholesterol absorption, and fermented red rice, a nutritional that reduce the synthesis of cholesterol. Subjects with sub optimal blood cholesterol levels, matching all the inclusion criteria and none of the exclusion criteria, will be treated for 8 weeks with a nutraceutical combination of phytosterols and fermented red rice and will have to maintain, during the entire duration of the study, the Mediterranean-style diet provided. The study will evaluate as primary objective the changes in LDL cholesterol blood levels and more in general the modulation of lipid profile and of others clinical parameters as well as the tolerability.

DETAILED DESCRIPTION:
The study is made up of four visits distributed over a 10-weeks period:

V 1 (day -14) - Screening: After providing written informed consent, tests will be run in order to check the subject's eligibility for the study. Subjects will also be given suggestions regarding their diet (a Mediterranean-style diet is to be maintained for the entire duration of the study).

V2 (baseline) and Day 0 (randomization): After confirmation of the subject's eligibility [LDL-C and Triglycerides (TG) criteria confirmed with blood test results], eligible subjects will be randomized within 3 days to one of the two treatment groups. During this visit an endothelial reactivity test will be performed.

V3 (28 ±3 days after Day 0) - Intermediate: Blood will be drawn for tests and compliance with treatment will be assessed. V4 (28 ± 3 days after Visit 3) - End of study: Blood tests and an endothelial reactivity test will be performed and treatment compliance will be assessed.

Weight, waist circumference, Index of Central Obesity (ICO) and Body Mass Index (BMI), Hepatic Steatosis Index (HSI) and Lipid Accumulation Product (LAP) will be measured/calculated at each visit, height at Visit 1.

Heart rate and blood pressure will be measured at each visit. Adverse events (AEs) will be collected throughout the study starting from the Informed consent signature.

The study will be monitored according to the details specified in the Monitoring Plan. The monitor will have the responsibility of reviewing the ongoing study with the Investigator to verify adherence to the protocol and to deal with any problems. Case Report Form (CRF) will be checked for completeness and consistency with the source data and special attention will be dedicated to patient enrolment, obtaining signed informed consent, occurrence of AEs, product accountability, and accurate recording of variables. The confidentiality of study related documents shall be maintained at all times. The Investigator agrees to allow access to all study materials needed for the proper review of study conduct.

An independent quality audit/inspection at the study site may take place at any time during or after the study. The independent audit/inspection can be carried out by the Sponsor's independent Quality Assurance (QA), by a Health Authorities or an Ethics Committee (EC).

ELIGIBILITY:
Inclusion Criteria:

-

Subjects must meet all of the following inclusion criteria:

* Age 30-75 years
* LDL-cholesterol = 115 -190 mg/dL
* Triglycerides < 400 mg/dL
* Any cardiovascular therapy should be stable for type and dose for at least three months
* Signed, written informed consent

Exclusion Criteria:

-

Subjects must meet none of the following exclusion criteria:

* Intolerance to any ingredient of dietary supplement
* Patients already suffering from cardiovascular diseases or at high risk of developing cardiovascular diseases
* Myopathies
* Uncontrolled diabetes mellitus based on PI judgment
* Chronic renal failure [defined as estimated glomerular filtration rate (eGFR) <60ml/min/1.73m2] or liver failure [defined as aspartate aminotransferase (AST) and /or Alanine Aminotransferase (ALT) >3 upper limit of normal (ULN)]
* Body Mass Index > 32 kg/m2
* Therapy with statins or other drugs or supplements with effects on lipid metabolism
* Patients with acquired immunodeficiency
* Treatment with immunosuppressants
* Pregnant or breastfeeding women
* Women of childbearing potential not willing to use effective birth control methods
* Patients participating or having participated in another clinical trial within the previous 3 months
* Current or recent history of drug or alcohol addiction based on PI judgment

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, Professor, Principal Investigator — Policlinico S.Orsola - Malpighi Medicina Interna Borghi
Locations (1):
- Policlinico S.Orsola - Malpighi Medicina Interna Borghi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cicero AFG, D'Addato S, Borghi C. A Randomized, Double-Blinded, Placebo-Controlled, Clinical Study of the Effects of a Nutraceutical Combination (LEVELIP DUO(R)) on LDL Cholesterol Levels and Lipid Pattern in Subjects with Sub-Optimal Blood Cholesterol Levels (NATCOL Study). Nutrients. 2020 Oct 14;12(10):3127. doi: 10.3390/nu12103127. PMID 33066334

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nutraceutical Combination | Placebo
Started | 44 | 44
Completed | 43 | 42
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population analysed is the Full Analysis Set one (FAS), composed by all randomization subjects who completed all the visits and were assessed for LDL cholesterol at last visit (Visit 4 - Week 8).
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutraceutical Combination | Placebo | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.28 (9.56) | 51.79 (10.74) | 51.53 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 43 | 42 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 43 | 42 | 85
LDL blood cholesterol level [Mean (Standard Deviation); unit: mg/dL] | 154.27 (20.47) | 160.57 (20.84) | 157.38 (20.77)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood LDL Cholesterol Level
Description: Mean change in blood LDL cholesterol level from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | -32.48 (30.18) | 2.54 (19.44)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean difference = -39.16, 95% CI 2-sided [-48.57 to -29.75]

2. Secondary Outcome: Change in Total Blood Cholesterol Level
Description: Mean change in total blood LDL cholesterol level from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | -31.99 (34.05) | 7.17 (21.10)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA; Least Square Mean difference = -41.24, 95% CI 2-sided [-51.73 to -30.74]

3. Secondary Outcome: Change in Blood HDL Cholesterol Level
Description: Mean change in blood HDL cholesterol level from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | 0.78 (7.17) | 1.11 (7.37)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.9510, ANCOVA; Least Square Mean difference = 0.09, 95% CI 2-sided [-2.87 to 3.05]

4. Secondary Outcome: Change in Blood Non-HDL Cholesterol Level
Description: Mean change in blood non-HDL cholesterol level from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | -33.35 (22.99) | 3.65 (18.78)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean difference = -41.70, 95% CI 2-sided [-51.58 to -31.82]

5. Secondary Outcome: Change in Blood Triglycerides Level
Description: Mean change in blood triglycerides level from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | -1.44 (42.76) | 17.62 (60.48)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.1924, ANCOVA; Least Square Mean difference = -7.00, 95% CI 2-sided [-17.59 to 3.59]

6. Secondary Outcome: Change in Blood Apolipoprotein B Level
Description: Mean change in blood apolipoprotein B level from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | -14.79 (15.05) | 1.6 (14.29)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean difference = -17.26, 95% CI 2-sided [-23.54 to -10.98]

7. Secondary Outcome: Change in Total Cholesterol/HDL Cholesterol Ratio
Description: Mean change in total cholesterol/HDL cholesterol ratio from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
ratio | -0.79 (0.79) | 0.06 (0.64)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean difference = -0.91, 95% CI 2-sided [-1.19 to -0.62]

8. Secondary Outcome: Change in Total LDL Cholesterol/HDL Cholesterol Ratio
Description: Mean change in LDL/HDL cholesterol ratio from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
ratio | -0.76 (0.70) | -0.01 (0.52)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean difference = -0.82, 95% CI 2-sided [-1.05 to -0.59]

9. Secondary Outcome: Change in Pulse Volume (PV) Waveform (Endothelial Reactivity)
Description: Mean change in Pulse Volume (PV) waveform from randomization (day 0) to V4 (week 8).
  PV unit of measurement is a percent change in the PV waveform area, comparing waveforms during and before hyperemia through the equation √PV2/PV1 that relates PV at baseline (PV1) and PV during hyperemia (PV2).
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
percentage of change | -0.08 (0.25) | -0.03 (0.21)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.4535, ANCOVA; Least Square Mean difference = -3.47, 95% CI 2-sided [-12.64 to 5.7]

10. Secondary Outcome: Change in Glycemia
Description: Mean change in Glycemia from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | -0.88 (6.26) | -1.57 (5.78)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.5594, ANCOVA; Least Square Mean difference = 0.74, 95% CI 2-sided [-1.76 to 3.24]

11. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: Mean change in aspartate aminotransferase from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
U/L | 0.98 (4.01) | 0.86 (3.40)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.9266, ANCOVA; Least Square Mean difference = -0.07, 95% CI 2-sided [-1.63 to 1.48]

12. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: Mean change in aspartate aminotransferase from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
U/L | 4.53 (9.29) | 2.93 (9.75)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.2654, ANCOVA; Least Square Mean difference = 6.02, 95% CI 2-sided [-4.66 to 16.69]

13. Secondary Outcome: Change in Gamma Glutamyl Transpeptidase (GGT)
Description: Mean change gamma glutamyl transpeptidase (GGT) from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
U/L | 0.91 (9.83) | 3.07 (9.53)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.2595, ANCOVA; Least Square Mean difference = -5.95, 95% CI 2-sided [-16.37 to 4.47]

14. Secondary Outcome: Change in Serum Creatinine
Description: Mean change in Serum Creatinine values from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | 0 (0.08) | 0 (0.10)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.8476, ANCOVA; Least Square Mean difference = 0.003, 95% CI 2-sided [-0.039 to 0.032]

15. Secondary Outcome: Change in Serum Uric Acid
Description: Mean change in Serum uric acid values from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
mg/dL | -0.30 (0.98) | 0 (0.56)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.1499, ANCOVA; Least Square Mean difference = -0.21, 95% CI 2-sided [-0.49 to 0.08]

16. Secondary Outcome: Change in Creatine Phosphokinase (CPK)
Description: Mean change in creatine phosphokinase (CPK) from randomization (day 0) to V4 (week 8)
Time Frame: From randomization (day 0) to V4 (week 8) for a total of 56 +/- 3 days of treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nutraceutical Combination | Placebo
Number analyzed (Participants) | 43 | 42
U/L | 2.09 (48.76) | -7.00 (56.56)
Statistical Analysis 1: Comparison: Nutraceutical Combination vs Placebo; Test type: Superiority; p = 0.7224, ANCOVA; Least Square Mean difference = 1.71, 95% CI 2-sided [-7.83 to 11.25]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from signature of the Informed Consent at screening visit, to the last visit (Visit 4) occurred 56 +/- 3 days after. Total period of AE collection throughout the study was of eleven months.
Arm/Group | Nutraceutical Combination | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

LIMITATIONS AND CAVEATS:
No limitations or caveats are applicable to this summary

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03739242/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT03739242/SAP_001.pdf